CLINICAL TRIAL: NCT06122740
Title: Reliability and Validity Studies of Turkish Version of Manual Ability Measure-36 (MAM-36)
Brief Title: Reliability and Validity Studies of Turkish Version of Manual Ability Measure-36
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gulser CINBAZ, PhD(c), Istanbul Medeniyet University
Other Study IDs: 2663-GOA
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Multiple Sclerosis; Stroke; Upper Extremity Problem
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish Validity and Reliability of The MAM-36 Scale — The aim of this study is to adapt the Manual Ability Measure-36 (MAM-36) scale to Turkish society and to make its validity and reliability in Turkish.

SUMMARY:
This study aim was to investigate the validity and reliability of Turkish version of Manual Ability Measure-36 (MAM-36) in patients with neurological disease.

DETAILED DESCRIPTION:
The reliability and validity of the scale were initiated by language equivalence and cultural adaptation. The MAM-36 scale was translated into Turkish by two experienced physiotherapists who are native Turkish speakers and have a good command of English, following the translation procedures. The two translations were compared with each other and a single Turkish draft was created. This draft was translated back into English by two translators who are native English speakers and have a good command of Turkish. The two back translations were compared to each other and converted into a single form. The resulting form was compared with the original form and the final back-translation scale was created. All translation formats of the scale were examined in detail by those who translated the scale into Turkish and a jury consisting of experienced physiotherapists. At the end of the meeting, the pilot study form of the scale was created. The created draft was applied to 30 healthy individuals as a pilot study. The final version of the scale was created by evaluating the feedback obtained. The clinical phase of the study was carried out on 250 volunteer individuals who applied to Dokuz Eylül University Hospital Neurology Department Polyclinics and were diagnosed with MS, Parkinson's disease, and stroke, and who had various degrees of problems in hand dexterity and functions due to their diseases. To evaluate the validity of MAM-36, Disability of Arm Shoulder and Hand (DASH), which can measure manual dexterity and was validated in Turkish, was used. The scales were repeated 15 days later to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with a neurological disease (Stroke, Parkinson's or MS)
* At least one upper extremity is affected
* Being conscious enough to complete the survey and knowing how to read and write
* Agreeing to participate in the research
* Being over 18 years old

Exclusion Criteria:

* Having an upper extremity operation within the last 6 months
* Having had an attack or seizure in the last month
* Participating in any physical therapy program during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who were diagnosed with stroke, Parkinson's or Multiple Sclerosis and had problems with manual dexterity in at least one upper extremity were included in the study.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Manual Ability Measure-36 | baseline
  Manual Ability Measure-36 was used to measure hand functions. The scale is a task- and patient-oriented measurement tool. Scale items consist of tasks that are frequently performed in daily life. In the survey where individuals subjectively evaluate their manual skills, a 4-point Likert rating scale is used, where 1 is 'I cannot do', 2 is 'very difficult', 3 is 'somewhat difficult', 4 is 'easy'. As a result of this 4-grade scoring of the scale, each patient receives a score between 0-144 from the test. However, in order to facilitate the analysis of future studies on the scale, a 100-point conversion table was created by the creators of the test.
Disability of Arm Shoulder and Hand | baseline
  Disability of Arm Shoulder and Hand (DASH) was developed by the 'Institute of Work and Health Ontario and American Academy of Orthopedic Surgeons' for use in patients with upper extremity problems. DASH is a self-report scale that measures activity and participation limitations and level of disability in upper extremity disorders. The patient's symptoms and daily life activities are examined on a scale consisting of thirty questions. Grading of the scale is done with a Likert scale. For each task, the patient gives a difficulty rating between 1 and 5. These five difficulty levels are defined as 1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not at all. A score between 0-100 (0 = no apology, 100 = maximum apology) is obtained from the scale. A high score also indicates high functional disability. The scale has a Turkish cultural adaptation.

IPD SHARING:
Plan to Share IPD: No